CLINICAL TRIAL: NCT01623843
Title: Femoroacetabular Impingement RandomiSed Controlled Trial (FIRST); Sub-study: Femoroacetabular Impingement RandomiSed Controlled Trial With an Embedded Prospective Cohort (FIRST-EPIC)
Brief Title: Femoroacetabular Impingement RandomiSed Controlled Trial
Acronym: FIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McMaster Surgical Associates (Other); Canadian Orthopaedic Foundation (Other); American Orthopaedic Society for Sports Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIRST-01
Record Dates: First submitted 2012-06-17; First posted 2012-06-20 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Femoroacetabular Impingement
Keywords: FAI; randomized; hip arthroscopy; lavage; osteochondroplasty
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arthroscopic Lavage (Active Comparator): Participants have three hip portals (antero-lateral, mid anterior, distal antero-lateral) with limited capsulotomy allowing for a complete assessment of the central and peripheral compartments. The participant has a diagnostic arthroscopy and lavage of the hip joint with three litres of normal saline. No osteochondroplasty or rim resection is completed in this group. No instruments are used to treat minor cartilage or labral damage. The labrum should only be repaired if mechanically unstable once probed with visible displacement or chondrolabral separation. The labrum will be refixated only if the above criteria for labral instability is met.
  Interventions: Procedure: Arthroscopic Lavage
- Arthroscopic Osteochondroplasty (Experimental): After establishing standard portals, an inter-portal capsulotomy will be completed to allow for complete evaluation of the central compartment of the hip. Significant and obvious labral tears and cartilage damage will be addressed. The labrum will be repaired if mechanically unstable once probed with visible displacement or chondrolabral separation. The acetabular rim will be evaluated and any evident Pincer lesion will be resected using an arthroscopic burr under fluoroscopic guidance. Following this resection, the labrum will be refixated only if the criteria for labral instability is met. Following this, a limited capsulotomy will be completed along the head-neck junction of the femoral neck to allow for visualization and treatment of the impingement lesion in the peripheral compartment. For the FIRST-EPIC sub-study, participants will receive the osteochondroplasty intervention as per standard of care.
  Interventions: Procedure: Arthroscopic Osteochondroplasty

INTERVENTIONS:
Procedure: Arthroscopic Lavage — Lavage: inflammation debris caused from continual friction in the hip is washed out.
  Arms: Arthroscopic Lavage
Procedure: Arthroscopic Osteochondroplasty — Osteochondroplasty: reshaping the hip ball and socket ("osteoplasty" or "rim trimming").
  Arms: Arthroscopic Osteochondroplasty

SUMMARY:
The purpose of this study is to determine whether surgical correction of hip impingement morphology via arthroscopic osteochondroplasty (shaving of bone) will provide improved clinical results (decreased pain and improved function) in adult patients with femoroacetabular impingement (FAI) compared to arthroscopic lavage (washing out of painful inflammation debris) and treating obvious damage of the hip joint.

DETAILED DESCRIPTION:
Femoroacetabular impingement (FAI) is a condition of the hip where there is a mismatch of the ball and socket in the hip joint. This mismatch creates abnormal contact in the hip which can cause patients to experience hip pain. This can eventually lead to hip damage and osteoarthritis. Hip arthroscopy, a form of minimally invasive surgery has become a popular treatment option. The investigators are conducting a definitive randomized controlled trial (RCT) to determine whether surgical correction of the impingement morphology via arthroscopic osteochondroplasty (shaving of bone) will provide improved clinical results (decreased pain and improved function) in adult FAI patients compared to arthroscopic lavage (washing out of painful inflammation debris) and treating obvious damage of the hip joint.

Like most RCTs, FIRST is designed to demonstrate efficacy (i.e. that an intervention can work theoretically under optimal conditions). In order to address generalizability and improve external validity of the FIRST trial, we are including an external validation cohort using a "RCT with and Embedded ProspectIve Cohort design" (FIRST-EPIC). This pragmatic cohort will allow us to: 1) safeguard against bias attributable to patients declining to take part in the RCT; 2) corroborate or refute whether our efficacy (RCT) population represents the best case scenario (i.e. those with optimal response to osteochondroplasty); 3) evaluate effectiveness of osteochondroplasty and other standard of care treatments for FAI in patients with potentially distinct prognostic factors; and 4) evaluate the cost-effectiveness of the interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women ages 18 to 50 years
2. Hip pain for greater than 6 months with no relief from non-operative means (physiotherapy, non-steroidal anti-inflammatory medication, rest)
3. Documentation of failed physiotherapy, including core conditioning of the hip, back, and abdomen
4. CAM or Mixed Type FAI as diagnosed on x-rays and magnetic resonance imaging (MRI) or magnetic resonance arthrogram (MRA)
5. Temporary relief from an intra-articular hip injection
6. Informed consent from participant
7. Ability to speak, understand and read in the language of the clinical site

Exclusion Criteria:

1. Previous inclusion in a study involving FAI
2. Evidence of hip dysplasia (centre edge angle less than 20)
3. Presence of advanced hip osteoarthritis (Tonnis Grade 2 or 3)
4. Presence of other hip syndromes (concurrent non-FAI related pathology)
5. Previous trauma to the affected hip
6. Previous surgery on the affected hip or contralateral hip
7. Severe acetabular deformities (e.g. acetabular protrusion, coxa profunda, circumferential labral ossification)
8. Immunosuppressive medication use
9. Chronic pain syndromes
10. Significant medical co-morbidities (requiring daily assistance for ADLs)
11. History of paediatric hip disease (Legg-Calve-Perthes; slipped capital femoral epiphysis)
12. Ongoing litigation or compensation claims secondary to hip problems
13. Any other reasons given to exclude the patient

    * If a patient does not meet the eligibility criteria for the FIRST trial, they may be considered eligible for the FIRST-EPIC sub-study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Pain (measured using a Visual Analog Scale) | 12 months
  The VAS is one of the most frequently used pain rating scales in clinical practice and research. The VAS is a validated unidimensional scale that is easy to use, requires no verbal or reading skills, and is sufficiently versatile to be employed in a variety of settings. The VAS will be administered during routine follow up visits at baseline, 2 weeks, 6 weeks, 3 months, 6 months, and 12 months.

SECONDARY OUTCOMES:
Function (measured using the Hip Outcome Score) | 12 months
  The HOS is a self-administered hip score that was designed to capture hip function and outcomes following surgical therapies such as arthroscopy. The HOS has been shown to have the greatest clinimetric evidence for use in patients with FAI or labral tears.
Health-related quality of life (measured using the Short-Form 12) | 12 months
  The SF-12 may be self or interview-administered and will help document general health status as well as the burden of illness that FAI presents.
Function and lifestyle (measured using the International Hip Outcome Tool) | 12 months
  The iHOT-12 is a shorter version of the iHOT-33 designed to be easier to complete in routine clinical practice to measure both health-related quality of life and changes after treatment in young, active patients with hip disorders. This questionnaire has been shown to be valid, reliable, and responsive to change.
Health utility (measured using the Euro-Quol 5 Dimensions) | 12 months
  The EQ-5D is a standardized instrument for use as a measure of health outcome. The EQ-5D comprises five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The EQ-5D has been used in previous studies involving patients with hip pain and has been extensively validated. Our decision to the use EQ-5D was based upon our interest in collecting health utility data for a formal economic analysis.
Urinary function (measured using the Male/Female Lower Urinary Tract Symptoms questionnaires) | 12 months
  The two validated questionnaires selected that pertain to male and female urinary symptoms are gender specific variations of the International Consultation on Continence Questionnaire (ICIQ). The ICIQ-MLUTS (male) and ICIQ-FLUTS (female). These are validated patient-completed questionnaires, which evaluate male and female lower urinary tract symptoms (LUTS), as well as quality of life. Both questionnaires have demonstrated validity, reliability and responsiveness internally and externally.
Sexual function (measured using the International Index of Erectile Dysfunction and the Female Sexual Function Index) | 12 months
  The FSFI is a brief psychometrically sound and reliable tool that assesses female sexual function, and has proven ability to discriminate between clinical and nonclinical populations.The FSFI is also designed to measure the impact on quality of life. The IIEF is a brief self-administered questionnaire assessing sexual experience within the previous 4 weeks, consisting of 15 questions designed to address 5 relevant aspects of male sexual function, specifically erectile function, sexual desire, orgasmic function, intercourse satisfaction and overall satisfaction. This instrument is psychometrically sound with high sensitivity and specificity, which has been validated for administration in research and clinical settings, and across cultures with linguistically validated versions.
Complications / Adverse events | 12 and 24 months
  Includes additional surgery, infection, reduced range of motion, and other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Olufemi Ayeni, MD, MSc, FRCSC, Principal Investigator — McMaster Univerity
Locations (10):
- Canada (7):
  - Dalhousie University, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Fowler Kennedy Sports Medicine Clinic, London, Ontario
  - London Health Sciences, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - CHU de Québec, L'Hôtel-Dieu de Québec, Québec, Quebec
- Odense University Hospital, Odense, Denmark
- Finland (2):
  - Hatanpää Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganz R, Parvizi J, Beck M, Leunig M, Notzli H, Siebenrock KA. Femoroacetabular impingement: a cause for osteoarthritis of the hip. Clin Orthop Relat Res. 2003 Dec;(417):112-20. doi: 10.1097/01.blo.0000096804.78689.c2. PMID 14646708
- [Background] Lincoln M, Johnston K, Muldoon M, Santore R. Combined arthroscopic and modified open approach for cam femoroacetabular impingement: a preliminary experience. Arthroscopy. 2009 Apr;25(4):392-9. doi: 10.1016/j.arthro.2008.12.002. PMID 19341926
- [Background] Philippon MJ, Stubbs AJ, Schenker ML, Maxwell RB, Ganz R, Leunig M. Arthroscopic management of femoroacetabular impingement: osteoplasty technique and literature review. Am J Sports Med. 2007 Sep;35(9):1571-80. doi: 10.1177/0363546507300258. Epub 2007 Apr 9. PMID 17420508
- [Background] Larson CM, Giveans MR. Arthroscopic management of femoroacetabular impingement: early outcomes measures. Arthroscopy. 2008 May;24(5):540-6. doi: 10.1016/j.arthro.2007.11.007. Epub 2008 Jan 7. PMID 18442686
- [Background] Ng VY, Arora N, Best TM, Pan X, Ellis TJ. Efficacy of surgery for femoroacetabular impingement: a systematic review. Am J Sports Med. 2010 Nov;38(11):2337-45. doi: 10.1177/0363546510365530. Epub 2010 May 20. PMID 20489213
- [Background] Botser IB, Smith TW Jr, Nasser R, Domb BG. Open surgical dislocation versus arthroscopy for femoroacetabular impingement: a comparison of clinical outcomes. Arthroscopy. 2011 Feb;27(2):270-8. doi: 10.1016/j.arthro.2010.11.008. PMID 21266277
- [Background] Bedi A, Chen N, Robertson W, Kelly BT. The management of labral tears and femoroacetabular impingement of the hip in the young, active patient. Arthroscopy. 2008 Oct;24(10):1135-45. doi: 10.1016/j.arthro.2008.06.001. PMID 19028166
- [Background] Clohisy JC, Carlisle JC, Beaule PE, Kim YJ, Trousdale RT, Sierra RJ, Leunig M, Schoenecker PL, Millis MB. A systematic approach to the plain radiographic evaluation of the young adult hip. J Bone Joint Surg Am. 2008 Nov;90 Suppl 4(Suppl 4):47-66. doi: 10.2106/JBJS.H.00756. No abstract available. PMID 18984718
- [Background] Tannast M, Siebenrock KA, Anderson SE. Femoroacetabular impingement: radiographic diagnosis--what the radiologist should know. AJR Am J Roentgenol. 2007 Jun;188(6):1540-52. doi: 10.2214/AJR.06.0921. PMID 17515374
- [Background] Anderson SE, Siebenrock KA, Mamisch TC, Tannast M. Femoroacetabular impingement magnetic resonance imaging. Top Magn Reson Imaging. 2009 Jun;20(3):123-8. doi: 10.1097/RMR.0b013e3181d99459. PMID 20410801
- [Background] Notzli HP, Wyss TF, Stoecklin CH, Schmid MR, Treiber K, Hodler J. The contour of the femoral head-neck junction as a predictor for the risk of anterior impingement. J Bone Joint Surg Br. 2002 May;84(4):556-60. doi: 10.1302/0301-620x.84b4.12014. PMID 12043778
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Christensen CP, Althausen PL, Mittleman MA, Lee JA, McCarthy JC. The nonarthritic hip score: reliable and validated. Clin Orthop Relat Res. 2003 Jan;(406):75-83. doi: 10.1097/01.blo.0000043047.84315.4b. PMID 12579003
- [Background] Schenker ML, Martin R, Weiland DE, Philippon MJ. Current trends in hip arthroscopy: a review of injury diagnosis, techniques and outcome scoring. Current opinion in orthopeadics.2005;16:89-94.
- [Background] Thorborg K, Roos EM, Bartels EM, Petersen J, Holmich P. Validity, reliability and responsiveness of patient-reported outcome questionnaires when assessing hip and groin disability: a systematic review. Br J Sports Med. 2010 Dec;44(16):1186-96. doi: 10.1136/bjsm.2009.060889. Epub 2009 Aug 6. PMID 19666629
- [Background] Lodhia P, Slobogean GP, Noonan VK, Gilbart MK. Patient-reported outcome instruments for femoroacetabular impingement and hip labral pathology: a systematic review of the clinimetric evidence. Arthroscopy. 2011 Feb;27(2):279-86. doi: 10.1016/j.arthro.2010.08.002. Epub 2010 Oct 29. PMID 21035994
- [Derived] Kay J, Simunovic N, Ayeni OR; FIRST Investigators; Bhandari M, Bedi A, Jarvinen T, Musahl V, Naudie D, Seppanen M, Slobogean G, Thabane L, Duong A, Skelly M, Shanmugaraj A, Crouch S, Sprague S, Heels-Ansdell D, Buckingham L, Ramsay T, Lee J, Kousa P, Carsen S, Choudur H, Sim Y, Johnston K, Wong I, Murphy R, Sparavalo S, Whelan D, Khan R, Wood GCA, Howells F, Grant H, Zomar B, Pollock M, Willits K, Firth A, Wanlin S, Remtulla A, Kaniki N, Belzile EL, Turmel S, Jorgensen U, Gam-Pedersen A, Sihvonen R, Raivio Sihvonen M, Toivonen Sihvonen P, Pirjetta Routapohja M. Effect of Osteochondroplasty on Time to Reoperation After Arthroscopic Management of Femoroacetabular Impingement: Analysis of a Randomized Controlled Trial. Orthop J Sports Med. 2022 Apr 5;10(4):23259671211041400. doi: 10.1177/23259671211041400. eCollection 2022 Apr. PMID 35400136
- [Derived] Femoroacetabular Impingement Randomized Controlled Trial (FIRST) Investigators; Ayeni OR, Karlsson J, Heels-Ansdell D, Thabane L, Musahl V, Simunovic N, Duong A, Bhandari M, Bedi A, Jarvinen T, Naudie D, Seppanen M, Slobogean G, Skelly M, Shanmugaraj A, Crouch S, Sprague S, Buckingham L, Ramsay T, Lee J, Kousa P, Carsen S, Choudur H, Sim Y, Johnston K, Sprague S, Wong I, Murphy R, Sparavalo S, Whelan D, Khan R, Wood GCA, Howells F, Grant H, Naudie D, Zomar B, Pollock M, Willits K, Firth A, Wanlin S, Remtulla A, Kaniki N, Belzile EL, Turmel S, Jorgensen U, Gam-Pedersen A, Hatanpaa T, Sihvonen R, Raivio M, Toivonen P, Routapohja MP. Osteochondroplasty and Labral Repair for the Treatment of Young Adults With Femoroacetabular Impingement: A Randomized Controlled Trial. Am J Sports Med. 2021 Jan;49(1):25-34. doi: 10.1177/0363546520952804. Epub 2020 Sep 24. PMID 32970955
- [Derived] Simunovic N, Heels-Ansdell D, Thabane L, Ayeni OR; FIRST Investigators. Femoroacetabular Impingement Randomised controlled Trial (FIRST) - a multi-centre randomized controlled trial comparing arthroscopic lavage and arthroscopic osteochondroplasty on patient important outcomes and quality of life in the treatment of young adult (18-50 years) femoroacetabular impingement: a statistical analysis plan. Trials. 2018 Oct 29;19(1):588. doi: 10.1186/s13063-018-2965-0. PMID 30373659
- [Derived] FIRST Investigators. A multi-centre randomized controlled trial comparing arthroscopic osteochondroplasty and lavage with arthroscopic lavage alone on patient important outcomes and quality of life in the treatment of young adult (18-50) femoroacetabular impingement. BMC Musculoskelet Disord. 2015 Mar 20;16:64. doi: 10.1186/s12891-015-0500-y. PMID 25886958